CLINICAL TRIAL: NCT07190716
Title: A Randomized, Double-Blind, Placebo-Controlled Phase I Clinical Trial Evaluating the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Preliminary Pharmacodynamic Characteristics of a Single Dose of GR2301 Injection in Healthy Adult Subjects in China.
Brief Title: A Study to Evaluate the Safety of GR2301 Injection in Healthy Volunteers.
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genrix (Shanghai) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GR2301-001
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Single Ascending Dose; Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- GR2301 injection 1 (Experimental): GR2301 injection dose 1/Placebo，Subcutaneous
  Interventions: Biological: GR2301 injection
- GR2301 injection 2 (Experimental): GR2301 injection dose 2/Placebo，Subcutaneous
  Interventions: Biological: GR2301 injection
- GR2301 injection 3 (Experimental): GR2301 injection dose 3/Placebo，Subcutaneous
  Interventions: Biological: GR2301 injection
- GR2301 injection 4 (Experimental): GR2301 injection dose 4/Placebo，Subcutaneous
  Interventions: Biological: GR2301 injection
- GR2301 injection 5 (Experimental): GR2301 injection dose 5/Placebo，Subcutaneous
  Interventions: Biological: GR2301 injection

INTERVENTIONS:
Biological: GR2301 injection — IL15 monoclonal antibody

SUMMARY:
This is a randomized, double-blind, placebo-controlled Phase I clinical trial evaluating the safety, tolerability, pharmacokinetics, immunogenicity, and preliminary pharmacodynamic characteristics of GR2301 injection in healthy adult subjects in China.The GR2301 injection dosage will be gradually increased. All healthy subjects will receive a single subcutaneous injection. Following administration, subjects will be followed for at least 16 weeks ± 7 days.

ELIGIBILITY:
Main Inclusion Criteria:

1. BMI 19.0-28.0 kg/m², with male subjects weighing ≥50.0 kg and female subjects weighing ≥45.0 kg；
2. Understand and comply with the requirements of the clinical protocol, voluntarily participate in the clinical trial, and sign the informed consent form.

Main Exclusion Criteria:

1. A history of past or current conditions involving the nervous system, cardiovascular system, urinary system, digestive system, respiratory system, endocrine system, metabolic system, or other clearly documented medical conditions, which the investigator deems may pose a risk to the subject's safety or interfere with the conduct, progress, or completion of the trial.
2. History of drug use or substance abuse, or positive urine drug screening prior to enrollment.
3. Pregnant and breastfeeding women.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-10 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | up to week16
  Incidence of AEs

SECONDARY OUTCOMES:
Pharmacokinetics parameters | up to week16
  concentration of GR2301
Incidence of ADA. | up to week16

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality, China